CLINICAL TRIAL: NCT01115790
Title: A Phase 1 Study of LY2606368 in Patients With Advanced Cancer
Brief Title: A Phase 1 Study in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13129; I4D-MC-JTJA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-28; First posted 2010-05-04 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Advanced Cancer; Squamous Cell Carcinoma; Carcinoma, Squamous Cell of Head and Neck; Lung Squamous Cell Carcinoma Stage IV; Anal Squamous Cell Carcinoma; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prexasertib (Experimental)
  Interventions: Drug: Prexasertib

INTERVENTIONS:
Drug: Prexasertib — Prexasertib IV on day 1 of a 14 day cycle. The expected duration is 3 cycles (2 weeks each for a total of 6 weeks). Participants receiving clinical benefit may remain on study until disease progression, unacceptable toxicity or other criteria for discontinuation are met.
  Other Names: LY2606368

SUMMARY:
The primary purpose of Parts A and B of this study is to evaluate the safety and toxicity of prexasertib (an inhibitor of checkpoint kinase 1[chk 1]) in participants with advanced or metastatic cancer (Part A), or squamous cell cancer of the head and neck or squamous cell cancer of any tumor type (Part B). Part C of the study will evaluate prexasertib in three different groups of participants; those with squamous cell cancer of the head and neck that has recurred or spread to other parts of the body, those with squamous non-small cell lung cancer that has recurred or spread, and those with squamous cell cancer of the anus that is not curable by existing therapy.

DETAILED DESCRIPTION:
Part C added per protocol amendment (February, 2013).

ELIGIBILITY:
Inclusion Criteria:

* Must be appropriate candidate for experimental therapy, as determined by investigator, after available standard therapies have failed
* Have adequate organ function
* Prior Therapies: Systemic treatments: must have discontinued previous systemic treatments for cancer and recovered from the acute effects of therapy. Participants must have discontinued mitomycin-C or nitrosourea therapy at least 42 days and have discontinued any cytotoxic therapies at least 28 days prior to study enrollment. Radiation therapy and surgery: must be completed at least 4 weeks before study enrollment
* Part A: Must have diagnosis of cancer that is advanced or metastatic
* Part B: Must have histologically confirmed squamous cell cancer of the head and neck or must have squamous cell cancer of any tumor type
* Part C: Must have histological diagnosis of squamous cell cancer of the head and neck, histological or cytological diagnosis of squamous non-small-cell lung cancer, or histological diagnosis of Stage IIIB (N2 or N3) or Stage IV squamous cell cancer of the anus that is not curable by local therapy
* Must be available during the duration of the study and willing to follow the study procedures
* If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for three months following the last dose of study drug
* If the participant is a female of childbearing potential, must have had a negative serum or urine pregnancy test within 7 days of the first dose of study drug and must not be breast feeding

Exclusion Criteria:

* Must not have taken an unapproved drug as treatment for any indication within the last 28 days prior to starting study treatment
* Must not have an active symptomatic fungal, bacterial or viral infection, including human immunodeficiency virus (HIV) or Hepatitis A, B, or C
* Must not have a serious heart condition, such as congestive heart failure, unstable angina pectoris, or heart attack within the last three months
* Must not have systolic blood pressure <90 millimeters of mercury (mmHg) or recurrent symptomatic orthostatic hypotension
* Must not have a family history of long QTc syndrome or be taking drugs known to cause QTc prolongation or Torsades de Pointes
* Must not have a serotonin-secreting carcinoid tumor or a prior history of drug-induced serotonin syndrome
* Must not have acute leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Determination of a Recommended Phase 2 Dosing Regimen: Maximum Tolerated Dose (Parts A and B) | Time of first dose until last dose (estimated as up to 156 weeks)
Determination of Clinically Significant Safety Effects (Parts A and B) | Time of first dose until last dose (estimated as up to 156 weeks)
Percentage of Participants With a Complete or Partial Response (Overall Response Rate) (Part C) | Baseline until disease progression or death from any cause (estimated as up to 24 weeks)

SECONDARY OUTCOMES:
Percentage of Participants with Complete Response, Partial Response, or Stable Disease (Disease Control Rate) (Parts A, B, and C) | Baseline until disease progression or death from any cause (estimated as up to 24 weeks)
Progression Free Survival (Parts B and C) | Baseline to measured progressive disease (estimated up to 24 weeks)
Duration of Response (Parts B and C) | First observation of complete response (CR), partial response (PR), or stable disease (SD) to first observation of progressive disease or death (estimated up to 24 weeks)
Preliminary Pharmacokinetics of Prexasertib (Cmax) (Parts A, B, and C) | During Cycles 1 and 2
Preliminary Pharmacokinetics of Prexasertib (AUC) (Parts A, B, and C) | During Cycles 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Sarasota, Florida
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hong DS, Moore K, Patel M, Grant SC, Burris HA 3rd, William WN Jr, Jones S, Meric-Bernstam F, Infante J, Golden L, Zhang W, Martinez R, Wijayawardana S, Beckmann R, Lin AB, Eng C, Bendell J. Evaluation of Prexasertib, a Checkpoint Kinase 1 Inhibitor, in a Phase Ib Study of Patients with Squamous Cell Carcinoma. Clin Cancer Res. 2018 Jul 15;24(14):3263-3272. doi: 10.1158/1078-0432.CCR-17-3347. Epub 2018 Apr 11. PMID 29643063
- [Derived] Hong D, Infante J, Janku F, Jones S, Nguyen LM, Burris H, Naing A, Bauer TM, Piha-Paul S, Johnson FM, Kurzrock R, Golden L, Hynes S, Lin J, Lin AB, Bendell J. Phase I Study of LY2606368, a Checkpoint Kinase 1 Inhibitor, in Patients With Advanced Cancer. J Clin Oncol. 2016 May 20;34(15):1764-71. doi: 10.1200/JCO.2015.64.5788. Epub 2016 Apr 4. PMID 27044938